CLINICAL TRIAL: NCT00641732
Title: A Phase 2, Randomized, Active Comparator-Controlled, Dose-Ranging Study to Evaluate the Efficacy and Safety of TAK-442 in Subjects Undergoing Total Knee Replacement
Brief Title: Efficacy and Safety of TAK-442 in Subjects Undergoing Total Knee Replacement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TAK-442_201; U1111-1115-9359 (Registry Identifier: WHO)
Record Dates: First submitted 2008-03-18; First posted 2008-03-24 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-03

CONDITIONS: Venous Thromboembolism
Keywords: venous thromboembolism; oral anticoagulant; direct factor Xa inhibitor; total knee replacement; drug therapy
MeSH Terms: conditions — Venous Thromboembolism | interventions — 1-(1-(3-((6-chloronaphthalen-2-yl)sulfonyl)-2-hydroxypropanoyl)piperidin-4-yl)tetrahydropyrimidin-2(1H)-one; Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- TAK-442 40 mg QD (Experimental)
  Interventions: Drug: TAK-442
- TAK-442 80 mg QD (Experimental)
  Interventions: Drug: TAK-442
- TAK-442 10 mg BID (Experimental)
  Interventions: Drug: TAK-442
- TAK-442 20 mg BID (Experimental)
  Interventions: Drug: TAK-442
- TAK-442 40 mg BID (Experimental)
  Interventions: Drug: TAK-442
- TAK-442 80 mg BID (Experimental)
  Interventions: Drug: TAK-442
- Enoxaparin 30 mg BID (Active Comparator)
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: TAK-442 — TAK-442 40 mg, tablets, orally, once daily for up to 10 days.
  Arms: TAK-442 40 mg QD
Drug: TAK-442 — TAK-442 80 mg, tablets, orally, once daily for up to 10 days.
  Arms: TAK-442 80 mg QD
Drug: TAK-442 — TAK-442 10 mg, tablets, orally, twice daily for up to 10 days.
  Arms: TAK-442 10 mg BID
Drug: TAK-442 — TAK-442 20 mg, tablets, orally, twice daily for up to 10 days.
  Arms: TAK-442 20 mg BID
Drug: TAK-442 — TAK-442 40mg, tablets, orally, twice daily for up to 10 days.
  Arms: TAK-442 40 mg BID
Drug: TAK-442 — TAK-442 80 mg, tablets, orally, twice daily for up to 10 days.
  Arms: TAK-442 80 mg BID
Drug: Enoxaparin — Enoxaparin 30 mg, syringe, subcutaneous injection, twice daily for up to 10 days.
  Arms: Enoxaparin 30 mg BID

SUMMARY:
The purpose of this study is to determine if TAK-442, once daily (QD) or twice daily (BID), is as safe and effective as enoxaparin in preventing the development of blood clots after knee replacement surgery.

DETAILED DESCRIPTION:
Takeda Global Research & Development Center, Inc. is developing the compound TAK-442 as a candidate for the secondary prevention of atherothrombotic events in patients with acute coronary syndromes. TAK-442 is an oral inhibitor of activated factor X within the blood coagulation cascade.

Due to its critical role in propagating the coagulation cascade, activated factor X is now considered to be a therapeutic aim in the development of anticoagulant drugs. Therefore activated factor X inhibitors, are among the agents under investigation as treatments for the spectrum of thromboembolic diseases involving either the arterial or the venous system.

Short term anticoagulation is often used for the prevention of venous thromboembolism. Patients undergoing major orthopedic surgery are at particularly high risk of venous thromboembolism after surgery. Consequently, such patients are routinely given anticoagulant medication after surgery. Although parenteral (injectable) drugs, such as enoxaparin or fondaparinux, can be used for this indication, the need for subcutaneous injection is problematic once patients are discharged from hospital. With the push for shorter hospital stays, this issue is of increasing concern. Therefore, there is a need for new oral anticoagulants. Although warfarin can be used for out of hospital prophylaxis, the need for coagulation monitoring and dose adjustments complicates its use. The new oral anticoagulants have the potential to overcome this problem because they can be given in fixed doses without the need for coagulation monitoring.

The purpose of the current study is to evaluate the antithrombotic effect of TAK-442 in patients undergoing elective total knee replacement surgery. This study will be the first TAK-442 trial in patients.

Individuals who want to participate in this study will be required to provide written informed consent. Study participation is anticipated to be approximately 2.25 months. Multiple procedures will occur at each visit which may include fasting, blood collection, urine collection, physical examinations, electrocardiograms and bilateral venogram. Outside of the study center, participants randomized to enoxaparin will be required to administer study medication subcutaneously with a syringe.

ELIGIBILITY:
Inclusion Criteria

* Scheduled to undergo elective, unilateral, primary, total knee replacement.
* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
* Screening laboratory tests (including clinical chemistry, hematology, and complete urinalysis) are within the reference range for the testing laboratory or are determined not to compromise subject safety by the investigator.

Exclusion Criteria

* Received TAK-442 in a previous clinical study or as a therapeutic agent.
* Body weight greater than 150 kg.
* Known bleeding diathesis (including Von Willebrand's disease or Hemophilia A or B).
* History of intracerebral, intraocular, or gastrointestinal bleeding, or active gastric or duodenal ulceration, within the 6 months prior to Randomization.
* Is required to take or continues taking any disallowed medication, prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including throughout the treatment period of the study due to an increased risk of bleeding, and should be stopped at least 5 days prior to surgery and in accordance with the product information:

  * Parenteral anticoagulants
  * Unfractionated heparin
  * Low molecular weight heparin (eg, dalteparin, non-study enoxaparin)
  * Direct thrombin inhibitors (eg, bivalirudin, argatroban)
  * Factor Xa inhibitors (eg, fondaparinux)
  * Oral anticoagulants
  * Warfarin
  * Anisindione
  * Antiplatelet drugs
  * Aspirin greater than 162 mg/day
  * Clopidogrel
  * Ticlopidine
  * Cilostazol
  * Dipyridamole
  * Glycoprotein IIb/IIIa inhibitors (eg, abciximab, eptifibatide)
  * NSAIDs with a half life greater than or equal to 17 hours
  * Meloxicam
  * Fibrinolytic agents
  * tPA (alteplase, reteplase, tenecteplase)
* History of major surgery within 3 months prior to randomization; or deep vein thrombosis, pulmonary embolism, myocardial infarction, cerebrovascular accident, or transient ischemic attack within 6 months prior to randomization.
* History of hypersensitivity or allergies to other activated factor X inhibitors or enoxaparin (or other low molecular weight heparins).
* Condition prohibiting bilateral venography.
* Has had multiple or traumatic epidural or spinal punctures immediately prior to randomization (defined as grossly bloody or greater than 3 attempted cannulations).
* Requires use of an indwelling epidural catheter for post-operative analgesia.
* Severe hypertension defined as systolic blood pressure greater than 180 mmHg or diastolic blood pressure greater than 110 mmHg at Screening.
* Moderate to severe renal dysfunction or disease (based on calculated creatinine clearance less than 45 mL/min/1.73 m2) at Screening.
* Alanine aminotransferase level greater than 2.0 times the upper limit of normal, active liver disease, or jaundice at Screening.
* Anemia (hemoglobin less than 10.0 g per dL) or thrombocytopenia (platelet count less than 100 times 103 per uL) at screening.
* Taking aspirin greater than 162 mg per day.
* Abuses drugs (defined as any illicit drug use) or alcohol.
* History of cancer that has not been in remission for at least 5 years prior to the first dose of study drug. (This criterion does not include those subjects with basal cell or Stage 1 squamous cell carcinoma of the skin.)
* Currently participating in another investigational study or has participated in an investigational study within 30 days prior to Screening.
* Any other serious disease or condition at Screening or Randomization that would compromise subject safety or make it difficult to successfully manage and follow the subject according to the protocol.
* Requires the use of pneumatic compression post-operatively.
* Known inherited thrombophilic disorder such as the factor V Leiden or prothrombin gene mutations or deficiencies of antithrombin, protein C, or protein S.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1045 (Actual)
Dates: Start 2007-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Composite evaluation of All-Cause Mortality, Symptomatic and Asymptomatic Deep Vein Thrombosis and Symptomatic Pulmonary Embolism. | Day 10.
Incidence of Major Bleeding. | Day 10.

SECONDARY OUTCOMES:
Evaluation of Major Venous Thromboembolism (composite of Symptomatic or Asymptomatic Proximal Deep Vein Thrombosis, Symptomatic Objectively Confirmed Pulmonary Embolism, and Venous Thromboembolism-Related Death). | Day 10.
Evaluation of Symptomatic Venous Thromboembolism. | Day 10.
Evaluation of Proximal Deep Vein Thrombosis. | Day 10.
Evaluation of Distal Deep Vein Thrombosis. | Day 10.
Evaluation of clinically significant Non-Major Bleeding events. | Day 10.
Evaluation of Minor Bleeding events. | Day 10.

CONTACTS AND LOCATIONS:
Overall Officials: Executive Medical Director Clinical Science, Study Director — Takeda
Locations (64):
- United States (38):
  - Birmingham, Alabama
  - Tuscaloosa, Alabama
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Bakersfield, California
  - Fountain Valley, California
  - Long Beach, California
  - Montclair, California
  - Oceanside, California
  - Vista, California
  - Yuba City, California
  - Aurora, Colorado
  - Centennial, Colorado
  - Denver, Colorado
  - Bay Pines, Florida
  - Clearwater, Florida
  - DeLand, Florida
  - Gulf Breeze, Florida
  - Hollywood, Florida
  - Pinellas Park, Florida
  - Tamarac, Florida
  - Atlanta, Georgia
  - Boise, Idaho
  - Meridian, Idaho
  - Springfield, Illinois
  - Towson, Maryland
  - Charlotte, North Carolina
  - Greensboro, North Carolina
  - Cincinnati, Ohio
  - Tulsa, Oklahoma
  - Altoona, Pennsylvania
  - Johnstown, Pennsylvania
  - Charleston, South Carolina
  - Dallas, Texas
  - Grapenne, Texas
  - Lubbock, Texas
  - San Antonio, Texas
  - Spokane, Washington
- Canada (26):
  - Edmonton, Alberta
  - Red Deer, Alberta
  - Kelowna, British Columbia
  - Winnipeg, Manitoba
  - Fredericton, New Brunswick
  - Saint John, New Brunswick
  - Dartmouth, Nova Scotia
  - Ajax, Ontario
  - Burlington, Ontario
  - Cambridge, Ontario
  - Chatham, Ontario
  - Greater Sudbury, Ontario
  - Guelph, Ontario
  - Kitchener, Ontario
  - Newmarket, Ontario
  - Niagra Falls, Ontario
  - Oakville, Ontario
  - Oshawa, Ontario
  - Ottawa, Ontario
  - Saint Catherines, Ontario
  - Sarnia, Ontario
  - Scarborough Village, Ontario
  - Thunder Bay, Ontario
  - Windsor, Ontario
  - Montreal, Quebec
  - Charlottetown

REFERENCES:
- [Result] Weitz JI, Cao C, Eriksson BI, Fisher W, Kupfer S, Raskob G, Spaeder J, Turpie AG. A dose-finding study with TAK-442, an oral factor Xa inhibitor, in patients undergoing elective total knee replacement surgery. Thromb Haemost. 2010 Dec;104(6):1150-7. doi: 10.1160/TH10-05-0273. Epub 2010 Sep 30. PMID 20886185